CLINICAL TRIAL: NCT04839809
Title: A Phase 1, Two-Part Study to Assess the Safety, Tolerability, and Pharmacokinetics of Single Ascending Doses of CC-92480; the Relative Bioavailability Among Two Formulations of CC 92480; and Food Effect on the Exposures of Two Formulations of CC 92480 in Healthy Adult Subjects
Brief Title: A Study to Assess Safety, Tolerability, and Pharmacokinetics of CC-92480 Formulations in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-92480-CP-003
Record Dates: First submitted 2021-04-07; First posted 2021-04-09 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: Healthy Volunteers
Keywords: Healthy Volunteers; CC-92480; Pharmacokinetics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- CC-92480-02 (Formulation A) with Placebo (Experimental): CC-92480-02 (Formulation A) or matching placebo to be administered orally under fasted conditions.
  Interventions: Drug: CC-92480; Other: Placebo
- CC-92480 (Formulation B)- fasted condition (Experimental): A single oral dose of CC-92480 (Formulation B) administered under fasted conditions.
  Interventions: Drug: CC-92480
- CC-92480-02 (Formulation A) - fasted condition (Experimental): A single oral dose of CC-92480-02 (Formulation A) administered under fasted conditions.
  Interventions: Drug: CC-92480
- CC-92480 (Formulation B) - Low-fat meal (Experimental): A single oral dose of CC-92480 (Formulation B) administered under fed conditions (low-fat meal).
  Interventions: Drug: CC-92480
- CC-92480-02 (Formulation A) - high-fat meal (Experimental): A single oral dose of CC-92480-02 (Formulation A) administered under fed conditions (high-fat meal).
  Interventions: Drug: CC-92480

INTERVENTIONS:
Drug: CC-92480 — Oral
Other: Placebo — Oral
  Arms: CC-92480-02 (Formulation A) with Placebo

SUMMARY:
This is a Phase 1 study that will be conducted in 2 parts. Participants may participate in 1 part only.

* Part 1 will be a randomized, double-blind, placebo-controlled, single ascending dose study to evaluate the safety, tolerability, and PK of CC-92480-02 (Formulation A) administered orally under fasted conditions in healthy adult participants.
* Part 2 will be a randomized, open-label, 2 × 4 crossover study (Periods 1, 2, 3, and 4) to evaluate the relative bioavailability (RBA) of Formulation A versus Formulation B under fasted conditions and explore safety, tolerability, and PK effects of food on Formulation A and Formulation B in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

Participants must satisfy the following criteria to be enrolled in the study:

1. Must understand and voluntarily sign a written informed consent form (ICF) prior to any study-related assessments/procedures being conducted.
2. Healthy adult female of nonchildbearing potential or male of any race, between 18 to 55 years of age (inclusive) at the time of signing the ICF, and in good health as determined by the screening history and Physical examination (PE).
3. Agrees to abide by the requirements and restrictions outlined in the CC-92480 Pregnancy Prevention Plan for Participants in Clinical Trials.
4. For males:

   a. Practice true abstinence (which must be reviewed on a monthly basis, as applicable) or agree to use a barrier contraception not made of natural (animal) membrane (eg, latex or polyurethane condoms are acceptable) when engaging in sexual activity with a female of childbearing potential (FCBP) while on study medication, and for at 3 months after the last dose of study medication even if he has undergone a successful vasectomy.
5. For females:

   Female participants must have been surgically sterilized (hysterectomy or bilateral oophorectomy; proper documentation required) at least 6 months before screening or be postmenopausal (defined as 24 months without menses before screening, with a serum follicle-stimulation hormone (FSH) level of > 40 IU/L at screening.
6. Must have a body mass index between 18 and 33 kg/m2 (inclusive) at the time of signing the ICF.
7. Clinical laboratory test results must be within the respective reference ranges; or if not, the results be clinically insignificant according to the Investigator's medical judgment.
8. Participant must agree and be willing to consume a standard high-fat meal (which may contain gluten), for Part 2 participants only.

Exclusion Criteria:

The presence of any of the following will exclude a participant from enrollment:

1. Female of childbearing potential, pregnant, or breastfeeding.
2. History of any clinically significant and relevant neurological, gastrointestinal (GI), renal, hepatic, cardiovascular, psychological, pulmonary, metabolic, endocrine, hematological, allergic disease, drug allergies, or other major disorders as determined by the Investigator.
3. History of severe (eg, anaphylactic, anaphylactoid, Stevens-Johnson, angioedematous) reaction to a drug, or adverse reactions to multiple drugs.
4. Use of any prescribed systemic or topical medication (including but not limited to analgesics, anesthetics, etc) within 28 days of the first dose administration.
5. Use of any nonprescribed systemic or topical medication (including vitamin/mineral supplements, and herbal medicines) within 14 days of the first dose administration.
6. Donation of blood or plasma within 8 weeks before the first dose administration to a blood bank or blood donation center.
7. History of drug abuse (as defined by the current version of the Diagnostic and Statistical Manual [DSM]) within 2 years before first dose administration, or positive drug screening test reflecting consumption of illicit drugs.
8. History of alcohol abuse (as defined by the current version of the DSM) within 2 years before first dose administration, or positive alcohol screen.
9. Known to have serum hepatitis or known to be a carrier of hepatitis B surface antigen (HBsAg) or hepatitis C antibody (HCV Ab), or have a reactive result to the test for human immunodeficiency virus (HIV) antibodies at screening.
10. Use of tobacco- or nicotine-containing products within 3 months prior to Day -1, as assessed by medical history and physical examination, or positive urine cotinine test at screening.
11. Vaccination within 30 days of first dose administration or plans to receive vaccination (live and attenuated) within 30 days after dosing.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-01-19 (Actual); Primary Completion 2021-10-08 (Actual); Study Completion 2021-10-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics- Cmax Part 1 | Up to 96 hours after dosing
  Maximum plasma concentration of drug
Pharmacokinetics- Tmax Part 1 | Up to 96 hours after dosing
  Time to maximum plasma concentration
Pharmacokinetics- AUC0-∞Part 1 | Up to 96 hours after dosing
  Area under the plasma concentration-time curve from time zero to infinity
Pharmacokinetics- AUC0-t Part1 | Up to 96 hours after dosing
  Area under the plasma concentration-time curve from time zero to the last observable concentration
Pharmacokinetics- t½ Part 1 | Up to 96 hours after dosing
  Terminal elimination half-life
Pharmacokinetics- CL/F Part 1 | Up to 96 hours after dosing
  Apparent total plasma clearance
Pharmacokinetics- Vz/F Part 1 | Up to 96 hours after dosing
  Apparent volume of distribution
Pharmacokinetics- tlag Part 1 | Up to 96 hours after dosing
  Lag time between time of administration and start of absorption
Pharmacokinetics- Cmax Part 2 | Up to 96 hours after dosing
  Maximum plasma concentration of drug
Pharmacokinetics- Ratio of Cmax (Formulation A/Formulation B) Part 2 | Up to 96 hours after dosing
  Ratio of maximum plasma concentration of drug
Pharmacokinetics- AUC0-∞ Part 2 | Up to 96 hours after dosing
  Area under the plasma concentration-time curve from time zero to infinity
Pharmacokinetics- Ratio of AUC0-∞ (Formulation A/Formulation B) Part 2 | Up to 96 hours after dosing
  Ratio of area under the plasma concentration-time curve from time zero to infinity
Pharmacokinetics- AUC0-t Part 2 | Up to 96 hours after dosing
  Area under the plasma concentration-time curve from time zero to the last observable concentration
Pharmacokinetics- AUC0-t (Formulation A/Formulation B) Part 2 | Up to 96 hours after dosing
  Area under the plasma concentration-time curve from time zero to the last observable concentration
Pharmacokinetics- Tmax Part 2 | Up to 96 hours after dosing
  Time to maximum plasma concentration
Pharmacokinetics- t½ Part 2 | Up to 96 hours after dosing
  Terminal elimination half-life
Pharmacokinetics- CL/F Part 2 | Up to 96 hours after dosing
  Apparent total plasma clearance
Pharmacokinetics- Vz/F Part 2 | Up to 96 hours after dosing
  Apparent volume of distribution
Pharmacokinetics- tlag Part 2 | Up to 96 hours after dosing
  Lag time between time of administration and start of absorption

SECONDARY OUTCOMES:
Pharmacokinetics- Cmax (high-fat meal) | Up to 96 hours after dosing
  Maximum plasma concentration of drug
Pharmacokinetics- Ratio (Fed/Fasted) of Cmax (high-fat meal) | Up to 96 hours after dosing
  Ratio of maximum plasma concentration of drug
Pharmacokinetics- AUC0-∞(high-fat meal) | Up to 96 hours after dosing
  Area under the plasma concentration-time curve from time zero to infinity
Pharmacokinetics- Ratio (Fed/Fasted) of AUC0-∞ (high-fat meal) | Up to 96 hours after dosing
  Ratio of area under the plasma concentration-time curve from time zero to infinity
Pharmacokinetics- AUC0-t (high-fat meal) | Up to 96 hours after dosing
  Area under the plasma concentration-time curve from time zero to the last observable concentration
Pharmacokinetics- Ratio (Fed/Fasted) of AUC0-t (high-fat meal) | Up to 96 hours after dosing
  Ratio of area under the plasma concentration-time curve from time zero to the last observable concentration
Pharmacokinetics- Tmax (high-fat meal) | Up to 96 hours after dosing
  Time to maximum plasma concentration
Pharmacokinetics- AUC0-24 (high-fat meal) | Up to 96 hours after dosing
  Area under the plasma concentration-time curve from time zero to 24 hours post dose
Pharmacokinetics- t½ (high-fat meal) | Up to 96 hours after dosing
  Terminal elimination half-life
Pharmacokinetics- CL/F (high-fat meal) | Up to 96 hours after dosing
  Apparent total plasma clearance
Pharmacokinetics- Vz/F (high-fat meal) | Up to 96 hours after dosing
  Apparent volume of distribution
Pharmacokinetics- tlag (high-fat meal) | Up to 96 hours after dosing
  Lag time between time of administration and start of absorption
Pharmacokinetics- Cmax (low-fat meal) | Up to 96 hours after dosing
  Maximum plasma concentration of drug
Pharmacokinetics- Ratio (Fed/Fasted) of Cmax (low-fat meal) | Up to 96 hours after dosing
  Ratio of maximum plasma concentration of drug
Pharmacokinetics- AUC0-∞(low-fat meal) | Up to 96 hours after dosing
  Area under the plasma concentration-time curve from time zero to infinity
Pharmacokinetics- Ratio (Fed/Fasted) of AUC0-∞(low-fat meal) | Up to 96 hours after dosing
  Ratio of area under the plasma concentration-time curve from time zero to infinity
Pharmacokinetics- AUC0-t (low-fat meal) | Up to 96 hours after dosing
  Area under the plasma concentration-time curve from time zero to the last observable concentration
Pharmacokinetics- Ratio (Fed/Fasted) of AUC0-t (low-fat meal) | Up to 96 hours after dosing
  Ratio of area under the plasma concentration-time curve from time zero to the last observable concentration
Pharmacokinetics- Tmax (low-fat meal) | Up to 96 hours after dosing
  Time to maximum plasma concentration
Pharmacokinetics- t½ (low-fat meal) | Up to 96 hours after dosing
  Terminal elimination half-life
Pharmacokinetics- CL/F (low-fat meal) | Up to 96 hours after dosing
  Apparent total plasma clearance
Pharmacokinetics- Vz/F (low-fat meal) | Up to 96 hours after dosing
  Apparent volume of distribution
Pharmacokinetics- tlag (low-fat meal) | Up to 96 hours after dosing
  Lag time between time of administration and start of absorption
Incidence of Adverse Events (AEs) | From enrollment until at least 28 days after completion of study treatment
  An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a participant during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the participant's health, including laboratory test values, regardless of etiology. Any worsening (ie, any clinically significant adverse change in the frequency or intensity of a preexisting condition) should be considered an AE.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- PPD Phase 1 Clinic, Austin, Texas, United States